CLINICAL TRIAL: NCT02644447
Title: The Safety and Efficacy Assessment of Human Umbilical Cord-derived Mesenchymal Stem Cells (HUC-MSCs) With Injectable Collagen Scaffold Transplantation in Woman With Premature Ovarian Failure (POF)
Brief Title: Transplantation of HUC-MSCs With Injectable Collagen Scaffold for POF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-POF/IGDB
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2015-12

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HUC-MSCs Transplantation (Experimental)
  Interventions: Biological: HUC-MSCs Transplantation
- HUC-MSCs with Injectable Collagen Scaffold Transplantation (Experimental)
  Interventions: Biological: HUC-MSCs with Injectable Collagen Scaffold Transplantation

INTERVENTIONS:
Biological: HUC-MSCs Transplantation — The patients with POF that will undergo bilateral ovaries injection of 10 million allogeneic HUC-MSCs.
  Arms: HUC-MSCs Transplantation
Biological: HUC-MSCs with Injectable Collagen Scaffold Transplantation — The patients with POF that will undergo bilateral ovaries injection of 10 million allogeneic HUC-MSCs with injectable collagen scaffold.
  Arms: HUC-MSCs with Injectable Collagen Scaffold Transplantation

SUMMARY:
Cellular therapies are rapidly progressing fields and have shown immense promise in the treatment of damaged ovarian function. The purpose of this study is to determine safety and efficacy of intra-ovarian injection of allogeneic HUC-MSCs with injectable collagen scaffold in women with Premature Ovarian Failure (POF) and to study the preliminary efficacy of HUC-MSCs with injectable collagen scaffold injection on ovarian function improvement.

DETAILED DESCRIPTION:
The purpose of this study was to explore the therapeutic potency of the HUC-MSCs with injectable collagen scaffold transvaginal injection for POF women. The serum of each patient was kept and sent for laboratory test before the surgery. HUC-MSCs were isolated and cultured in vitro and the biomarkers of HUC-MSCs were detected using Flow cytometry detection. The HUC-MSCs with injectable collagen scaffold were then injected directly into bilateral ovaries. The outcomes of patients were examined after the injection. The patients are monitored for signs of follicle growth and growing follicles are stimulated with exogenous hormones, followed by oocyte retrieval and In Vitro Fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Premature Ovarian Failure.
2. Patients show no response to drug treatment
3. Women between 20 and 39 years.
4. Willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Abnormal karyotyping (e.g. turner syndrome, fragile X syndrome).
2. Congenital ovarian malformation.
3. Severe endometriosis.
4. Thyroid dysfunction.
5. Contraindications for pregnancy.
6. Contraindications for hormone replacement therapy.
7. Prior personal history of ovarian cancer or after radiotherapy.
8. Unwilling to comply with follow-up schedule or want to take other treatment during the follow-up period.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by Adverse Events | Up to 6 months
  Proportion of patients with postoperative infections and serious adverse events (SAEs) were assessed by long term follow-up.

SECONDARY OUTCOMES:
Number of Antral follicle development | Once a week within 3 months after the surgery
  The number of follicles developing was recorded by transvaginal ultrasound scan.
Estradiol (E2) serum level | Once a week within 3 months after the surgery
  Serum E2 level was evaluated after surgery.
Follicle Stimulating Hormone (FSH) serum level | Once a week within 3 months after the surgery
  Serum FSH level was evaluated after surgery.
Anti-Mullerian Hormone (AMH) serum level | Once a week within 3 months after the surgery
  Serum AMH level was evelated after surgery.
Pregnancy rate | 2 weeks after embryo implantation
  The incidence of pregnancy following transfer of embryos produced from oocytes recovered from follicles developing was assessed by Serum Human Chorionic Gonadotropin (HCG) detection.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China